CLINICAL TRIAL: NCT03506490
Title: Acute Effects of Aerobic Exercise on Motor Memory Consolidation in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Castelo Branco (Other)
Responsible Party: Principal Investigator, André Ramalho, Principal Investigator, Instituto Politécnico de Castelo Branco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ESE IPCB03
Record Dates: First submitted 2018-04-14; First posted 2018-04-24 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Elderly
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): The participants of this study were 33 subjects of both genders (M = 68 years old; SD = 4.2 years old) and were divided in two groups: a control group (N = 15; M = 67, 6 years old; SD = 4.1 years old) and an experimental group (N = 18; M = 67, 4 years old; SD = 4.4 years old). The participants performed a Soda Pop test before the aerobic training session (Baseline). The training session lasted 45 minutes and was composed of running exercises. After the training session, the motor memory consolidation was held in three different stages: Training; 1 hour after training; 24 hours after training.
  Interventions: Other: Aerobic exercises

INTERVENTIONS:
Other: Aerobic exercises — The training session lasted 45 minutes and was composed of running exercises.

SUMMARY:
Scientific evidence suggests that an aerobic exercise session promotes improvements in the consolidation of motor memory in adults. In this sense, the main purpose of this study was to investigate if an aerobic training session could improve motor memory consolidation in older people.

DETAILED DESCRIPTION:
The participants of this study were 33 subjects of both genders (M = 68 years old; SD = 4.2 years old) and were divided in two groups: a control group (N = 15; M = 67, 6 years old; SD = 4.1 years old) and an experimental group (N = 18; M = 67, 4 years old; SD = 4.4 years old). The participants performed a Soda Pop test before the aerobic training session (Baseline). The training session lasted 45 minutes and was composed of running exercises. After the training session, the motor memory consolidation was held in three different stages: Training; 1 hour after training; 24 hours after training.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* sensory abnormalities;
* mental abnormalities;
* motor abnormalities;
* other atypical health problems.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — * individuals not engaged in physical activity;
  * persons aged from 65 years.
Enrollment: 33 (Actual)
Dates: Start 2013-01-03 (Actual); Primary Completion 2013-07-05 (Actual); Study Completion 2013-09-15 (Actual)

PRIMARY OUTCOMES:
The participants performed a Soda Pop test before the aerobic training session (Baseline). | The participants performed a Soda Pop test before the aerobic training session (Baseline).
  The participants performed a Soda Pop test before the aerobic training session (Baseline).